CLINICAL TRIAL: NCT02084719
Title: Comparison of OraQuick HCV Rapid Antibody Test and Standard Serologic Screening for Hepatitis C: Validity, Acceptability and Impact on Linkage to Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitement
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Valérie Martel-Laferrière, MD, MS, FRCPC, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 01
Record Dates: First submitted 2014-03-07; First posted 2014-03-12 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Active or Ex-injection Drug Users; Indication of Hepatitis C Screening
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Patients will be tests with both the standard algorithm and the Oraquick HCV Rapid Antibody Test
  Interventions: Device: Oraquick HCV Rapid Antibody Test; Device: Standard algorithm
- Group B (Active Comparator): Patients will be tested only with the standard algorithm
  Interventions: Device: Standard algorithm

INTERVENTIONS:
Device: Oraquick HCV Rapid Antibody Test
  Arms: Group A
Device: Standard algorithm

SUMMARY:
Rapid tests are increasingly used in medical practice, notably to screen for HIV. Their use has been associated with a faster linkage to care and lower rates of loss to follow up. Rapid tests are also well accepted by patients and clinicians.

No rapid test is currently approved in Canada for screening of hepatitis C. Hepatitis C diagnosis is done through based on blood testing and the screening algorithm may require up to 3 visits to clarify the hepatitis C status.

The Oraquick HCV test is a rapid test done on blood or saliva that can replace the first step of the regular screening algorithm. With this test the initial screening and the confirmation test can be done in one visit.

The primary endpoint of this pilot-project is to evaluate clinical characteristics of Oracquick HCV (sensitivity, specificity, positive and negative predictive values) and to compare them to those of the standard screening algorithm in a population of active or ex-users of injected drugs. The project also intend to evaluate if the rapid test can reduce the rates of loss to follow up and increase the linkage to hepatitis C specialized care. This last endpoint will be evaluated through phone call follow up 6 months after the screening.

One hundred and fifty patients will be included. Half will be tested with the standard algorithm and the Oraquick HCV test (group A) and half will be tested only with the standard algorithm.

Results of group A will be used to determine the clinical characteristics of Oraquick HCV. Results of groups A and B will be used to evaluate rates of loss to follow up, costs avoided by the use of the rapid test and linkage to care of infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Indication of hepatitis C screening
* Active or ex-injection drug user

Exclusion Criteria:

* Known hepatitis C infection
* Unknown HIV status and patient refusing to HIV testing

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients for whom Oraquick HCV Antibody Test accurately diagnosed anti-HCV status | Patients will be followed for an expected average of 6 weeks
  Oraquick HCV Antibody test will be compared to a composite goldstandard:
  * If both the Oraquick test and the standard test are negative, the results will be considered as a true negative.
  * If both the Oraquick test and the standard test are positive, the results will be considered as a true positive.
  * If the tests are discordant, HCV RNA testing will be performed. If HCV RNA is positive, the result of the test who predicted the positive result will be a true positive and the result of the other test will be a false negative. If the HCV RNA is negative, the result of the standard test will be considered as the true value (either positive or negative).

SECONDARY OUTCOMES:
Loss to follow up | 3 months
  Proportion of patients not completing the screening procedures
Linkage to care | 6 months
  Proportion of infected patients initiating a follow up with an hepatitis C specialized provider
Avoided costs | 6 months
  Costs that could have been avoided by the use of the rapid test.
Satisfaction | 15 minutes
  Patients and provider satisfaction about the test

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Martel-Laferrière, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada